CLINICAL TRIAL: NCT00741104
Title: A Feasibility Study Exploring the Effect of Remicade on the Disease Activity in RA Patients
Brief Title: A Feasibility Study Exploring the Effect of Remicade on the Disease Activity in RA Patients (Study P05417)
Acronym: REQUEST
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05417
Record Dates: First submitted 2008-07-30; First posted 2008-08-26 (Estimated); Results first posted 2009-08-21 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients: Patients on maintenance therapy for RA with infliximab for >= the past 12 months.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Treatment of RA with Infliximab according to and under normal routine clinical practice.
  Other Names: Remicade; SCH 215596

SUMMARY:
This observational study will explore the Swedish national population of patients with rheumatoid arthritis (RA) on infliximab maintenance therapy in order to identify patients who may be eligible for a dose reduction study. Patients will be asked a variety of questions regarding their treatment dosing and disease activity, and then asked whether or not they would consider participating in a dose reduction study. Patients in this study will be described in terms of demographic and disease characteristics.

DETAILED DESCRIPTION:
Already known Subjects (RA and on at least 12 months ongoing Remicade treatment) from the clinic could participate if they are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis, infliximab maintenance treatment for at least the past 12 months, given written informed consent.

Exclusion Criteria:

* episodic treatment with infliximab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are Swedish patients on maintenance therapy for RA with infliximab for >= the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

REFERENCES:
- [Result] Breynaert C, Ferrante M, Fidder H, Van Steen K, Noman M, Ballet V, Vermeire S, Rutgeerts P, Van Assche G. Tolerability of shortened infliximab infusion times in patients with inflammatory bowel diseases: a single-center cohort study. Am J Gastroenterol. 2011 Apr;106(4):778-85. doi: 10.1038/ajg.2011.61. Epub 2011 Mar 15. PMID 21407184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Information about patients' doctor visits prior to this study were obtained from the Swedish Rheumatology Register and the South Swedish Arthritis Treatment Group.
Pre-assignment Details: RA patients in Sweden normally see their doctor every 6 months. Information obtained from these visits are entered into national registries. Data in this study were based on retrospective review of the two visits preceding the study visit and the visit when infliximab was prescribed for the 1st time, as well as the one and only study visit.
Groups:
- RA Patients: Patients on maintenance therapy for rheumatoid arthritis (RA) with infliximab for >= the past 12 months.
Period: Overall Study
Arm/Group | RA Patients
Started | 363
Completed | 363
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RA Patients
Number analyzed (Participants) | 363
Age, Continuous [Mean (Full Range); unit: years] | 61 [23 to 89]
Gender [Count of Participants; unit: Participants]
  Female | 254
  Male | 109
Region of Enrollment [Number; unit: participants]
  Sweden | 363
Change in dosing interval since previous doctor visit [Number; unit: participants] — Only 264 patients had this information available from the registry databases.
  participants
    Decreased dosing interval | 19
    No change | 226
    Increased dosing interval | 19
    Data unavailable | 99

OUTCOME MEASURES:

1. Primary Outcome: Dosing Interval Between the Infliximab Infusions
Description: Patients were asked as part of the Remicade questionnaire what dosing interval they were on.
Time Frame: Measured from the Remicade Questionnaire at first (and only) study visit
Measure: Number; unit: participants
Arm/Group | RA Patients
Number analyzed (Participants) | 363
participants
  < every 8 weeks | 121
  every 8 weeks | 205
  > every 8 weeks | 37

2. Secondary Outcome: Disease Activity Score Based on Assessment of 28 Joints (DAS28), Health Assessment Questionnaire (HAQ), C-reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), Infliximab Dosage.
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed
Time Frame: Measured at first (and only) study visit, and outcomes measured during the two preceding physician visits are extracted from the Swedish Rheumatoid Arthritis (RA) Registry.
Reporting Status: Not Posted

3. Secondary Outcome: Adverse Events (AEs)
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed
Time Frame: Collected at first (and only) study visit, all AEs reported during the previous 12 months is collected from the Swedish Rheumatoid Arthritis (RA) Registry.
Reporting Status: Not Posted

4. Secondary Outcome: Duration of Subject's Rheumatoid Arthritis (RA) Diagnosis, European Quality of Life Group 1990 5 Dimension (EQ5D) and Patient Remicade Questionnaire.
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed
Time Frame: as for outcome 2
Reporting Status: Not Posted

5. Primary Outcome: Reason for Extending Dosing Interval
Description: Among patients who reported that they at some occasion during treatment with infliximab had a longer dosing interval than every 8 weeks, the reason for extending dosing interval was asked of each patient.
Time Frame: Measured from the Remicade Questionnaire at first (and only) study visit
Population: Among the 363 patients, 106 patients reported that they at SOME occasion during treatment with infliximab had had a longer dosing interval than every 8 weeks.
Measure: Number; unit: participants
Arm/Group | RA Patients
Number analyzed (Participants) | 106
participants
  decreased disease activity | 24
  doctor's advice | 31
  surgery/co-morbidity | 28
  vacation/stay abroad | 14
  pregnancy/trying to become pregnant | 0
  other | 9

6. Primary Outcome: Patient Response to Increased Dosing Interval
Description: Among patients who reported that they at some occasion during treatment with infliximab had a longer dosing interval than every 8 weeks, patients were asked "did you notice any difference when your dosing interval was extended?" Those who noticed a difference were asked if their experience was positive or negative.
Time Frame: Measured from the Remicade Questionnaire at first (and only) study visit
Population: Among the 363 patients, 106 patients reported that they at SOME occasion during treatment with infliximab had had a longer dosing interval than every 8 weeks. Among the 106 patients who increased dosing interval, 79 noticed a difference. These 79 were analyzed for this measure.
Measure: Number; unit: participants
Arm/Group | RA Patients
Number analyzed (Participants) | 79
participants
  positive | 4
  negative | 75

7. Primary Outcome: Number of Patients Agreeing to Participate in a Dose Reduction Study
Description: As part of the Remicade questionnaire, patients were asked "would you consider participating in a dose reduction study?"
Time Frame: Measured from the Remicade Questionnaire at first (and only) study visit
Population: Out of the 363 subjects in the analysis, 361 subjects answered this question.
Measure: Number; unit: participants
Arm/Group | RA Patients
Number analyzed (Participants) | 361
participants
  no | 139
  yes | 222

ADVERSE EVENTS:
Arm/Group | RA Patients
Serious Adverse Events (participants affected / at risk) | 0/363
Other Adverse Events (participants affected / at risk) | 0/363

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to publish/publicly present any interim results of the Study. PI further agrees to provide 45 days written notice to Sponsor prior to submission for publication/presentation to permit Sponsor to review drafts of any material before publication which report any results arising out of the Study. Sponsor shall have the right to review and comment.